CLINICAL TRIAL: NCT06773299
Title: ENhancing Intergenerational HeAlth in Nigeria: Peripartum as Critical Life StagE for CardioVascular Health
Acronym: ENHANCE-CVH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Abuja Teaching Hospital (Other); New York University (Other); Parents as Teachers (Unknown)
Responsible Party: Principal Investigator, Mark Huffman, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01HL168771 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2025-01-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Hypertension in Pregnancy; Hypertension; Obesity and Overweight; Maternal Morbidity and Mortality; Maternal and Child Health Outcomes
Keywords: Maternal Hypertension; Maternal and infant cardiovascular health; Hybrid Type 2 effectiveness-implementation; Obesity in pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Obesity; Overweight; Pregnancy in Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAT+HEALTH Intervention (Experimental): Participants randomized to this arm will receive 40 biweekly PAT+HEALTH intervention delivery ante- and postnatally. These will primarily focus on promoting cardiovascular health for mother and child through lifestyle and behavioral modifications along with additional support and education for pregnancy and cardiovascular health.
  Interventions: Behavioral: PAT+HEALTH curriculum - Nigeria
- Control (No Intervention): Participants randomized to the control group will not receive the PAT+HEALTH intervention and will only receive standard ante- and postnatal care.

INTERVENTIONS:
Behavioral: PAT+HEALTH curriculum - Nigeria — This intervention is an adaption of the PAT Curriculum and the HEALTH intervention specifically tailored for the Nigerian context.
  Arms: PAT+HEALTH Intervention

SUMMARY:
The purpose of the ENHANCE-CVH study is to promote intergenerational cardiovascular health (CVH) of women and children in Abuja and the surrounding Federal Capital Territory of Nigeria. The study team plans to achieve this through an adaptation of an existing evidence based intervention - Parents as Teachers (PAT) curriculum + Healthy Eating Active Living Taught at Home (HEALTH) - among pregnant women with obesity and their children in Nigeria. The aim of the study is to evaluate the effectiveness and implementation of community health educator-led delivery of the PAT+HEALTH intervention via home visits to answer the following main questions:

* Will the women participating in the intervention have a greater change in weight from baseline to 18-month follow up compared to the women who do not?
* Will the women and children in the intervention group display better CVH promoting lifestyle behaviors compared to those in the control group?

Participants in the study will complete baseline surveys and have clinical data, lab data, and body measurements captured. Participants will also have these procedures repeated at birth and every 6 months up to 24 months post-delivery. Once randomized to the intervention group, participants will complete 40 biweekly PAT+HEALTH curriculum delivery sessions, each lasting approximately 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

•≥18 years of age,

* Pregnant women under 14 weeks gestation,
* Singleton gestation,
* Body mass index > 30 kg/m2
* Willing to participate in ENHANCE CVH for 2 years,
* Planning to receive prenatal care and deliver at either one of the participating primary healthcare, centers or University of Abuja Teaching Hospital, and
* Able to give informed consent for study participation, understanding she and her child will both be involved.

Exclusion Criteria:

* Current enrollment in a weight loss program,
* Inability to engage in a walking program,
* Active substance abuse
* Treatment with medications known to impact weight (e.g., corticosteroids, antipsychotics),
* Plan to relocate within the next 2 years, or
* Unwilling to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in maternal body weight from baseline | Baseline to 18-month postnatal follow up
  Between group difference in change in maternal body weight f rom baseline to 18-month follow-up measured in kilograms.

SECONDARY OUTCOMES:
Change in cardiovascular health score | Baseline to 18-month postnatal follow up
  Between group difference in change in maternal cardiovascular health score (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Tobacco Use/Exposure | Baseline to 18-month postnatal follow up
  Between group difference in change in Tobacco Use/exposure subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Diet | Baseline to 18-month postnatal follow up
  Between group difference in change in Diet subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Physical Activity | Baseline to 18-month postnatal follow up
  Between group difference in change in Physical Activity subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - BMI | Baseline to 18-month postnatal follow up
  Between group difference in change in BMI subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Blood Pressure | Baseline to 18-month postnatal follow up
  Between group difference in change in blood pressure subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Cholesterol | Baseline to 18-month postnatal follow up
  Between group difference in change in cholesterol subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Blood Sugar | Baseline to 18-month postnatal follow up
  Between group difference in change in Blood Sugar subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in cardiovascular health score - Sleep | Baseline to 18-month postnatal follow up
  Between group difference in change in Sleep subscore (range from 0-100: Life's Essential 8) from baseline to 18-month postnatal follow-up.
Change in Child CVH behaviors - Diet | Birth to 18 months
  Between group difference in child cardiovascular health behaviors as measured through parent-reported diet from birth to 18 months.
Change in Child CVH behaviors - Physical Activity | Birth to 18 months
  Between group difference in child cardiovascular health behaviors as measured through parent-reported activity from birth to 18 months using the Movement Behavior Questionnaire - Child Open Version (MBQ-C)
Change in Child CVH behaviors - Sleep | Birth to 18 months
  Between group difference in child cardiovascular health behaviors as measured through parent-reported sleep from birth to 18 months using the Brief Infant Sleep Questionnaire - Revised version (BISQ-R)
Maternal Mortality | Baseline to 18-month postnatal follow up
  Between group difference in composite rate of maternal mortality from baseline to 18 months postnatal follow-up
Maternal morbidity | Baseline to 18-month postnatal follow up
  Between group difference in composite rate of maternal morbidity (defined as occurrence of any serious adverse event) from baseline to 18 month postnatal follow-up.
Stillbirth or spontaneous abortion | Measured at Birth
  Between group difference in the composite rate of stillbirth or spontaneous abortion.
Neonatal, infant, and child mortality | Birth to 18 months
  Between group difference in the composite rate of neonatal, infant, or childhood mortality from birth to 18 months.
Neonatal, infant, and child morbidity | Birth to 18 months
  Between group difference in the composite rate of neonatal, infant, or childhood morbidity as defined by occurrence of any serious adverse events from birth to 18 months.

OTHER OUTCOMES:
Child Weight for length | Birth, 6 months, 18 months
  Between group difference in child weight-for-length z-score at 6 and 18 months, adjusted for weight-for-length z-score at birth.
Child BMI | Birth, 6 months, 18 months
  Between group difference in child BMI z-score at 6 and 18 months, adjusted for weight-for-length z-score at birth.
Parental feeding behaviors | 6 months, 12 months, 18 months, 24 months
  Parental feeding behaviors measured by the Feeding to Manage Child Behavior Questionnaire (FMCBQ)

CONTACTS AND LOCATIONS:
Overall Officials: Dike B Ojji, MD, Principal Investigator — University of Abuja Teaching Hospital
Locations (1):
- University of Abuja Teaching Hospital, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available after the conclusion of the study following the guidelines of BioData Catalyst. A codebook will be provided.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning not later than 6 months after publication of results with no end date.
Access Criteria: Those who have privileges to access data stored within the BioData Catalyst repository may access the data as per the rules and regulations of that system. Data provided to BioData Catalyst will be completely de-identified following their criteria.

REFERENCES:
- [Background] GBD 2019 Demographics Collaborators. Global age-sex-specific fertility, mortality, healthy life expectancy (HALE), and population estimates in 204 countries and territories, 1950-2019: a comprehensive demographic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1160-1203. doi: 10.1016/S0140-6736(20)30977-6. PMID 33069325
- [Background] Tukur J, Lavin T, Adanikin A, Abdussalam M, Bankole K, Ekott MI, Godwin A, Ibrahim HA, Ikechukwu O, Kadas SA, Nwokeji-Onwe L, Nzeribe E, Ogunkunle TO, Oyeneyin L, Tunau KA, Bello M, Aminu I, Ezekwe B, Aboyeji P, Adesina OA, Chama C, Etuk S, Galadanci H, Ikechebelu J, Oladapo OT; Maternal and Perinatal Database for Quality, Equity and Dignity Network. Quality and outcomes of maternal and perinatal care for 76,563 pregnancies reported in a nationwide network of Nigerian referral-level hospitals. EClinicalMedicine. 2022 Apr 28;47:101411. doi: 10.1016/j.eclinm.2022.101411. eCollection 2022 May. PMID 35518118
- [Background] Abubakar I, Dalglish SL, Angell B, Sanuade O, Abimbola S, Adamu AL, Adetifa IMO, Colbourn T, Ogunlesi AO, Onwujekwe O, Owoaje ET, Okeke IN, Adeyemo A, Aliyu G, Aliyu MH, Aliyu SH, Ameh EA, Archibong B, Ezeh A, Gadanya MA, Ihekweazu C, Ihekweazu V, Iliyasu Z, Kwaku Chiroma A, Mabayoje DA, Nasir Sambo M, Obaro S, Yinka-Ogunleye A, Okonofua F, Oni T, Onyimadu O, Pate MA, Salako BL, Shuaib F, Tsiga-Ahmed F, Zanna FH. The Lancet Nigeria Commission: investing in health and the future of the nation. Lancet. 2022 Mar 19;399(10330):1155-1200. doi: 10.1016/S0140-6736(21)02488-0. Epub 2022 Mar 15. No abstract available. PMID 35303470
- [Background] Parikh NI, Gonzalez JM, Anderson CAM, Judd SE, Rexrode KM, Hlatky MA, Gunderson EP, Stuart JJ, Vaidya D; American Heart Association Council on Epidemiology and Prevention; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; and the Stroke Council. Adverse Pregnancy Outcomes and Cardiovascular Disease Risk: Unique Opportunities for Cardiovascular Disease Prevention in Women: A Scientific Statement From the American Heart Association. Circulation. 2021 May 4;143(18):e902-e916. doi: 10.1161/CIR.0000000000000961. Epub 2021 Mar 29. PMID 33779213
- [Background] Nigeria Federal Ministry of Health (2019). National Multi-Sectoral Action Plan for the Prevention and Control of Non-Communicable Diseases; Federal Capital Territory, Nigeria.
- [Background] Aifah A, Onakomaiya D, Iwelunmor J, Oladele D, Gbajabiamila T, Obiezu-Umeh C, Nwaozuru U, Musa AZ, Ezechi O, Ogedegbe G. Nurses' perceptions on implementing a task-shifting/sharing strategy for hypertension management in patients with HIV in Nigeria: a group concept mapping study. Implement Sci Commun. 2020 Jun 26;1:58. doi: 10.1186/s43058-020-00048-y. eCollection 2020. PMID 32885213
- [Background] Wiltsey Stirman S, Baumann AA, Miller CJ. The FRAME: an expanded framework for reporting adaptations and modifications to evidence-based interventions. Implement Sci. 2019 Jun 6;14(1):58. doi: 10.1186/s13012-019-0898-y. PMID 31171014
- [Background] Haire-Joshu D, Schwarz CD, Steger-May K, Lapka C, Schechtman K, Brownson RC, Tabak RG. A Randomized Trial of Weight Change in a National Home Visiting Program. Am J Prev Med. 2018 Mar;54(3):341-351. doi: 10.1016/j.amepre.2017.12.012. PMID 29455756
- [Background] Haire-Joshu D, Cahill AG, Stein RI, Cade WT, Woolfolk CL, Moley K, Mathur A, Schwarz CD, Schechtman KB, Klein S. Randomized Controlled Trial of Home-Based Lifestyle Therapy on Postpartum Weight in Underserved Women with Overweight or Obesity. Obesity (Silver Spring). 2019 Apr;27(4):535-541. doi: 10.1002/oby.22413. PMID 30900408
- [Background] Cahill AG, Haire-Joshu D, Cade WT, Stein RI, Woolfolk CL, Moley K, Mathur A, Schechtman K, Klein S. Weight Control Program and Gestational Weight Gain in Disadvantaged Women with Overweight or Obesity: A Randomized Clinical Trial. Obesity (Silver Spring). 2018 Mar;26(3):485-491. doi: 10.1002/oby.22070. PMID 29464907
- [Background] Ojji DB, Baldridge AS, Orji IA, Shedul GL, Ojo TM, Ye J, Chopra A, Ale BM, Shedul G, Ugwuneji EN, Egenti NB, Aluka-Omitiran K, Okoli RCB, Eze H, Nwankwo A, Banigbe B, Tripathi P, Kandula NR, Hirschhorn LR, Huffman MD; Hypertension Treatment in Nigeria Program Investigators. Characteristics, treatment, and control of hypertension in public primary healthcare centers in Nigeria: baseline results from the Hypertension Treatment in Nigeria Program. J Hypertens. 2022 May 1;40(5):888-896. doi: 10.1097/HJH.0000000000003089. Epub 2022 Jan 15. PMID 35034080
- [Background] Glasgow RE, Battaglia C, McCreight M, Ayele RA, Rabin BA. Making Implementation Science More Rapid: Use of the RE-AIM Framework for Mid-Course Adaptations Across Five Health Services Research Projects in the Veterans Health Administration. Front Public Health. 2020 May 27;8:194. doi: 10.3389/fpubh.2020.00194. eCollection 2020. PMID 32528921
- [Background] Gemechu KS, Assefa N, Mengistie B. Prevalence of hypertensive disorders of pregnancy and pregnancy outcomes in Sub-Saharan Africa: A systematic review and meta-analysis. Womens Health (Lond). 2020 Jan-Dec;16:1745506520973105. doi: 10.1177/1745506520973105. PMID 33334273
- [Background] Adeloye D, Ige-Elegbede JO, Ezejimofor M, Owolabi EO, Ezeigwe N, Omoyele C, Mpazanje RG, Dewan MT, Agogo E, Gadanya MA, Alemu W, Harhay MO, Auta A, Adebiyi AO. Estimating the prevalence of overweight and obesity in Nigeria in 2020: a systematic review and meta-analysis. Ann Med. 2021 Dec;53(1):495-507. doi: 10.1080/07853890.2021.1897665. PMID 33783281
- [Background] Institute of Medicine (US) and National Research Council (US) Committee to Reexamine IOM Pregnancy Weight Guidelines; Rasmussen KM, Yaktine AL, editors. Weight Gain During Pregnancy: Reexamining the Guidelines. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32813/ PMID 20669500
- [Background] Teede HJ, Bailey C, Moran LJ, Bahri Khomami M, Enticott J, Ranasinha S, Rogozinska E, Skouteris H, Boyle JA, Thangaratinam S, Harrison CL. Association of Antenatal Diet and Physical Activity-Based Interventions With Gestational Weight Gain and Pregnancy Outcomes: A Systematic Review and Meta-analysis. JAMA Intern Med. 2022 Feb 1;182(2):106-114. doi: 10.1001/jamainternmed.2021.6373. PMID 34928300
- [Background] Mandy M, Nyirenda M. Developmental Origins of Health and Disease: the relevance to developing nations. Int Health. 2018 Mar 1;10(2):66-70. doi: 10.1093/inthealth/ihy006. PMID 29528398
- [Background] Barker DJ. Fetal origins of coronary heart disease. BMJ. 1995 Jul 15;311(6998):171-4. doi: 10.1136/bmj.311.6998.171. PMID 7613432
- [Background] Jebasingh F, Thomas N. Barker Hypothesis and Hypertension. Front Public Health. 2022 Jan 21;9:767545. doi: 10.3389/fpubh.2021.767545. eCollection 2021. PMID 35127619
- [Background] Bhargava SK, Sachdev HS, Fall CH, Osmond C, Lakshmy R, Barker DJ, Biswas SK, Ramji S, Prabhakaran D, Reddy KS. Relation of serial changes in childhood body-mass index to impaired glucose tolerance in young adulthood. N Engl J Med. 2004 Feb 26;350(9):865-75. doi: 10.1056/NEJMoa035698. PMID 14985484
- [Background] Haire-Joshu D, Tabak R. Preventing Obesity Across Generations: Evidence for Early Life Intervention. Annu Rev Public Health. 2016;37:253-71. doi: 10.1146/annurev-publhealth-032315-021859. PMID 26989828
- [Background] Khalil A, Huffman MD, Prabhakaran D, Osmond C, Fall CH, Tandon N, Lakshmy R, Prabhakaran P, Biswas SK, Ramji S, Sachdev HS, Bhargava SK; New Delhi Birth Cohort. Predictors of carotid intima-media thickness and carotid plaque in young Indian adults: the New Delhi birth cohort. Int J Cardiol. 2013 Aug 20;167(4):1322-8. doi: 10.1016/j.ijcard.2012.03.180. Epub 2012 Apr 25. PMID 22537976
- [Background] Huffman MD, Khalil A, Osmond C, Fall CH, Tandon N, Lakshmy R, Ramji S, Gera T, Prabhakaran P, Dey Biswas SK, Reddy KS, Bhargava SK, Sachdev HS, Prabhakaran D; New Delhi Birth Cohort. Association between anthropometry, cardiometabolic risk factors, & early life factors & adult measures of endothelial function: Results from the New Delhi Birth Cohort. Indian J Med Res. 2015 Dec;142(6):690-8. doi: 10.4103/0971-5916.174559. PMID 26831418
- [Background] Paul IM, Savage JS, Anzman-Frasca S, Marini ME, Beiler JS, Hess LB, Loken E, Birch LL. Effect of a Responsive Parenting Educational Intervention on Childhood Weight Outcomes at 3 Years of Age: The INSIGHT Randomized Clinical Trial. JAMA. 2018 Aug 7;320(5):461-468. doi: 10.1001/jama.2018.9432. PMID 30088009
- [Background] Phelan S, Clifton RG, Haire-Joshu D, Redman LM, Van Horn L, Evans M, Joshipura K, Couch KA, Arteaga SS, Cahill AG, Drews KL, Franks PW, Gallagher D, Josefson JL, Klein S, Knowler WC, Martin CK, Peaceman AM, Thom EA, Wing RR, Yanovski SZ, Pi-Sunyer X; LIFE-Moms Research Group. One-year postpartum anthropometric outcomes in mothers and children in the LIFE-Moms lifestyle intervention clinical trials. Int J Obes (Lond). 2020 Jan;44(1):57-68. doi: 10.1038/s41366-019-0410-4. Epub 2019 Jul 10. PMID 31292531
- [Background] Leunissen RW, Kerkhof GF, Stijnen T, Hokken-Koelega A. Timing and tempo of first-year rapid growth in relation to cardiovascular and metabolic risk profile in early adulthood. JAMA. 2009 Jun 3;301(21):2234-42. doi: 10.1001/jama.2009.761. PMID 19491185
- [Background] Ong KK, Ahmed ML, Emmett PM, Preece MA, Dunger DB. Association between postnatal catch-up growth and obesity in childhood: prospective cohort study. BMJ. 2000 Apr 8;320(7240):967-71. doi: 10.1136/bmj.320.7240.967. PMID 10753147
- [Background] Sirard JR, Pate RR. Physical activity assessment in children and adolescents. Sports Med. 2001;31(6):439-54. doi: 10.2165/00007256-200131060-00004. PMID 11394563
- [Background] Tabak RG, Morshed AB, Schwarz CD, Haire-Joshu D. Weight gain prevention content delivered to mothers: Lessons from an intervention embedded in a community organization. Obes Sci Pract. 2019 Nov 18;5(6):540-547. doi: 10.1002/osp4.369. eCollection 2019 Dec. PMID 31890244
- [Background] Cole TJ, Power C, Moore GE. Intergenerational obesity involves both the father and the mother. Am J Clin Nutr. 2008 May;87(5):1535-6; author reply 1536-7. doi: 10.1093/ajcn/87.5.1535. No abstract available. PMID 18469281
- [Background] Sutherland G, Brown S, Yelland J. Applying a social disparities lens to obesity in pregnancy to inform efforts to intervene. Midwifery. 2013 Apr;29(4):338-43. doi: 10.1016/j.midw.2012.01.016. Epub 2012 Nov 9. PMID 23146141
- [Background] Wen LM, Baur LA, Simpson JM, Rissel C, Wardle K, Flood VM. Effectiveness of home based early intervention on children's BMI at age 2: randomised controlled trial. BMJ. 2012 Jun 26;344:e3732. doi: 10.1136/bmj.e3732. PMID 22735103
- [Background] Savage JS, Birch LL, Marini M, Anzman-Frasca S, Paul IM. Effect of the INSIGHT Responsive Parenting Intervention on Rapid Infant Weight Gain and Overweight Status at Age 1 Year: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):742-9. doi: 10.1001/jamapediatrics.2016.0445. PMID 27271455
- [Background] Seidler AL, Hunter KE, Johnson BJ, Ekambareshwar M, Taki S, Mauch CE, Mihrshahi S, Askie L, Campbell KJ, Daniels L, Taylor RW, Wen LM, Byrne R, Lawrence J, Perlstein R, Wardle K, Golley RK. Understanding, comparing and learning from the four EPOCH early childhood obesity prevention interventions: A multi-methods study. Pediatr Obes. 2020 Nov;15(11):e12679. doi: 10.1111/ijpo.12679. Epub 2020 Jun 15. PMID 32543054
- [Background] Phelan JC, Link BG, Tehranifar P. Social conditions as fundamental causes of health inequalities: theory, evidence, and policy implications. J Health Soc Behav. 2010;51 Suppl:S28-40. doi: 10.1177/0022146510383498. PMID 20943581
- [Background] Solar O, Irwin A. (2010) A Conceptual Framework for Action on the Social Determinants of Health. Social Determinants of Health Discussion Paper 2 (Policy and Practice). Geneva, Switzerland.
- [Background] National Population Commission (NPC) [Nigeria] and ICF. Nigeria Demographic and Health Survey (NDHS) 2018. Abuja, Nigeria, and Rockville, Maryland, USA: NPC and ICF.
- [Background] Adepoju P. Nigeria's new law aims to provide health insurance to all. Lancet. 2022 Jun 4;399(10341):2092. doi: 10.1016/S0140-6736(22)01008-X. No abstract available. PMID 35658984
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] Antenatal Care: An Orientation Package for Health Care Providers. (2017) Nigeria Federal Ministry of Health Guidelines. Federal Capital Territory, Nigeria.
- [Background] Ojji DB, Baldridge AS, Orji AI, Shedul LG, Ojji OI, Egenti NB, Nwankwo AM, Huffman MD. Feasibility and effect of community health worker support and home monitoring for blood pressure control in Nigeria: a randomised pilot trial. Cardiovasc J Afr. 2020 May-Jun;31(3):213-215. doi: 10.5830/CVJA-2019-066. PMID 32627803
- [Background] Baldridge AS, Aluka-Omitiran K, Orji IA, Shedul GL, Ojo TM, Eze H, Shedul G, Ugwuneji EN, Egenti NB, Okoli RCB, Ale BM, Nwankwo A, Osagie S, Ye J, Chopra A, Sanuade OA, Tripathi P, Kandula NR, Hirschhorn LR, Huffman MD, Ojji DB. Hypertension Treatment in Nigeria (HTN) Program: rationale and design for a type 2 hybrid, effectiveness, and implementation interrupted time series trial. Implement Sci Commun. 2022 Aug 2;3(1):84. doi: 10.1186/s43058-022-00328-9. PMID 35918703
- [Background] Ojji D, Aifah A, Dulli L, Iwelunmor J; MAP-IT Study Team. Early stakeholder engagement lessons from managing hypertension among people living with human-immunodeficiency virus: an integrated model (MAP-IT). Eur Heart J. 2022 Jul 1;43(25):2347-2349. doi: 10.1093/eurheartj/ehac159. No abstract available. PMID 35441679
- [Background] Ojji D; Nigeria Sodium Study Team. Developing long-term strategies to reduce excess salt consumption in Nigeria. Eur Heart J. 2022 Mar 31;43(13):1277-1279. doi: 10.1093/eurheartj/ehac025. No abstract available. PMID 35134903
- [Background] Dietary Guidelines Advisory Committee. 2020. Scientific Report of the 2020 Dietary Guidelines Advisory Committee: Advisory Report to the Secretary of Agriculture and the Secretary of Health and Human Services. U.S. Department of Agriculture, Agricultural Research Service, Washington, DC. Available at: Https://Doi.Org/10.52570/DGAC2020.
- [Background] Holtrop JS, Rabin BA, Glasgow RE. Qualitative approaches to use of the RE-AIM framework: rationale and methods. BMC Health Serv Res. 2018 Mar 13;18(1):177. doi: 10.1186/s12913-018-2938-8. PMID 29534729
- [Background] Shelton RC, Chambers DA, Glasgow RE. An Extension of RE-AIM to Enhance Sustainability: Addressing Dynamic Context and Promoting Health Equity Over Time. Front Public Health. 2020 May 12;8:134. doi: 10.3389/fpubh.2020.00134. eCollection 2020. PMID 32478025
- [Background] Gale RC, Wu J, Erhardt T, Bounthavong M, Reardon CM, Damschroder LJ, Midboe AM. Comparison of rapid vs in-depth qualitative analytic methods from a process evaluation of academic detailing in the Veterans Health Administration. Implement Sci. 2019 Feb 1;14(1):11. doi: 10.1186/s13012-019-0853-y. PMID 30709368
- [Background] Kirk MA, Moore JE, Wiltsey Stirman S, Birken SA. Towards a comprehensive model for understanding adaptations' impact: the model for adaptation design and impact (MADI). Implement Sci. 2020 Jul 20;15(1):56. doi: 10.1186/s13012-020-01021-y. PMID 32690104
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Orji IA, Baldridge AS, Omitiran K, Guo M, Ajisegiri WS, Ojo TM, Shedul G, Kandula NR, Hirschhorn LR, Huffman MD, Ojji DB. Capacity and site readiness for hypertension control program implementation in the Federal Capital Territory of Nigeria: a cross-sectional study. BMC Health Serv Res. 2021 Apr 9;21(1):322. doi: 10.1186/s12913-021-06320-8. PMID 33836719
- [Background] Huffman MD, Capewell S, Ning H, Shay CM, Ford ES, Lloyd-Jones DM. Cardiovascular health behavior and health factor changes (1988-2008) and projections to 2020: results from the National Health and Nutrition Examination Surveys. Circulation. 2012 May 29;125(21):2595-602. doi: 10.1161/CIRCULATIONAHA.111.070722. Epub 2012 Apr 30. PMID 22547667
- [Background] Riley L, Guthold R, Cowan M, Savin S, Bhatti L, Armstrong T, Bonita R. The World Health Organization STEPwise Approach to Noncommunicable Disease Risk-Factor Surveillance: Methods, Challenges, and Opportunities. Am J Public Health. 2016 Jan;106(1):74-8. doi: 10.2105/AJPH.2015.302962. PMID 26696288
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027
- [Background] American Academy of Pediatrics. Bright Futures: Prevention and Health Promotion for Infants, Children, Adolescents, and Their Families. 2021; Https://Brightfutures.Aap.Org/Pages/Default.Aspx. Accessed July 25, 2022.
- [Background] Kapp JM, Hall B, Kemner A. Collecting Early Childhood Obesity Measurements Through a Home Visiting Program: A Proof-of-Concept Study. Prev Chronic Dis. 2020 Dec 31;17:E169. doi: 10.5888/pcd17.200214. PMID 33416469
- [Background] Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of Obesity and Severe Obesity in US Children, 1999-2016. Pediatrics. 2018 Mar;141(3):e20173459. doi: 10.1542/peds.2017-3459. PMID 29483202
- [Background] O'Connor EA, Evans CV, Burda BU, Walsh ES, Eder M, Lozano P. Screening for Obesity and Intervention for Weight Management in Children and Adolescents: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2017 Jun 20;317(23):2427-2444. doi: 10.1001/jama.2017.0332. PMID 28632873
- [Background] WHO Child Growth Standards. Int J Pediatrics. 2006; 95(S450): 1-106. doi: 10.1080/08035320500495373
- [Background] Ebrahim GJ. WHO Child Growth Standards. Growth velocity based on weight, length and head circumference: methods and development. J Trop Pediatrics. 2010;56(2):136-136. doi:10.1093/tropej/fmp086
- [Background] Hamilton CM, Strader LC, Pratt JG, Maiese D, Hendershot T, Kwok RK, Hammond JA, Huggins W, Jackman D, Pan H, Nettles DS, Beaty TH, Farrer LA, Kraft P, Marazita ML, Ordovas JM, Pato CN, Spitz MR, Wagener D, Williams M, Junkins HA, Harlan WR, Ramos EM, Haines J. The PhenX Toolkit: get the most from your measures. Am J Epidemiol. 2011 Aug 1;174(3):253-60. doi: 10.1093/aje/kwr193. Epub 2011 Jul 11. PMID 21749974
- [Background] Thompson T, McQueen A, Croston M, Luke A, Caito N, Quinn K, Funaro J, Kreuter MW. Social Needs and Health-Related Outcomes Among Medicaid Beneficiaries. Health Educ Behav. 2019 Jun;46(3):436-444. doi: 10.1177/1090198118822724. Epub 2019 Jan 17. PMID 30654655
- [Background] Sullivan SD, Mauskopf JA, Augustovski F, Jaime Caro J, Lee KM, Minchin M, Orlewska E, Penna P, Rodriguez Barrios JM, Shau WY. Budget impact analysis-principles of good practice: report of the ISPOR 2012 Budget Impact Analysis Good Practice II Task Force. Value Health. 2014 Jan-Feb;17(1):5-14. doi: 10.1016/j.jval.2013.08.2291. Epub 2013 Dec 13. PMID 24438712
- [Background] Calhoun A, Mainor A, Moreland-Russell S, Maier RC, Brossart L, Luke DA. Using the Program Sustainability Assessment Tool to assess and plan for sustainability. Prev Chronic Dis. 2014 Jan 23;11:130185. doi: 10.5888/pcd11.130185. PMID 24456644
- [Background] Luke DA, Calhoun A, Robichaux CB, Elliott MB, Moreland-Russell S. The Program Sustainability Assessment Tool: a new instrument for public health programs. Prev Chronic Dis. 2014 Jan 23;11:130184. doi: 10.5888/pcd11.130184. PMID 24456645
- [Derived] Lopez JD, Aifah A, Nartey C, Ripiye NR, Shedul GL, Okpetu E, Nwaozuru UC, Aluka-Omitiran K, Onwu N, Obiezu-Umeh C, Marshall T, Kemner A, Lindley KJ, Haire-Joshu D, Davila-Roman VG, Akaba G, Huffman MD, Ojji DB, Okoro CE; ENHANCE C. V. H. Investigators. Enhancing intergenerational HeAlth in Nigeria: peripartum as Critical life stagE for CardioVascular Health (ENHANCE-CVH) study: findings from pre-implementation using the updated consolidated framework for implementation research (CFIR 2.0). Implement Sci Commun. 2025 Dec 4;7(1):5. doi: 10.1186/s43058-025-00816-8. PMID 41345984
- See also: Related Info — https://linkscommunity.org/assets/PDFs/nigeria-hypertension-protocol-04.pdf